CLINICAL TRIAL: NCT01099748
Title: Open Label, Single-Sequence Study To Estimate The Effect Of Lersivirine (UK-453,061) On S- And R-Methadone In Subjects Receiving Chronic Methadone Treatment
Brief Title: Estimate The Effect Of Lersivirine On The Pharmacokinetics Of S- And R-Methadone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A5271031
Record Dates: First submitted 2010-04-05; First posted 2010-04-07 (Estimated); Last update posted 2010-08-30 (Estimated); Status verified 2010-08

CONDITIONS: Healthy Volunteers
Keywords: Drug interaction; pharmacokinetics; lersivirine; methadone
MeSH Terms: interventions — Methadone; UK 453,061

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methadone (Active Comparator): Dose of methadone must not change from 1 week prior to study start and through the duration of the study.
  Interventions: Drug: Methadone
- Lersivirine + Methadone (Experimental)
  Interventions: Drug: Lersivirine + Methadone

INTERVENTIONS:
Drug: Methadone — Methadone 50 - 150 mg QD (Day 1)
  Arms: Methadone
Drug: Lersivirine + Methadone — Lersivirine 1000 mg QD + Methadone 50 - 150 mg QD (Days 2-11)
  Arms: Lersivirine + Methadone

SUMMARY:
The objective of this study is to estimate the effect of lersivirine on the pharmacokinetics of R-methadone and S-methadone and to investigate the safety and tolerability of lersivirine when co-administered with methadone. Symptoms of methadone withdrawal will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history except drug abuse), full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of 17.5 to 35.5 kg/m2; and a total body weight >50 kg (110 lbs).
* Receiving stable methadone maintenance treatment for at least 3 months (dose range 50-150 mg QD).

Exclusion Criteria:

* Subjects on therapy for Hepatitis B and/or Hepatitis C; Evidence of impaired liver function (ie, AST and/or ALT greater than 3 times the upper limit of normal, total bilirubin >1.5 times the upper limit of normal, albumin <3.5 g/dL).
* 12-lead ECG demonstrating QTc >450 msec for males and QTc >470 msec for females or any other clinically significant abnormalities at screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2010-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
R-methadone and S-methadone plasma pharmacokinetic parameters: AUC24, Cmax, Tmax, and C24h on Days 1 and 11 | Day 12

SECONDARY OUTCOMES:
Safety and toleration assessed by spontaneous reporting of adverse events, vital signs, 12-lead ECG and laboratory safety assessments | Day 12
Symptoms of methadone withdrawal as assessed by the Short Opiate Withdrawal Scale (SOWS), Desires for Drug Questionnaire (DDQ) and Pupillary Diameter measurement performed on Days 0 -12. | Day 12

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5271031&StudyName=Estimate%20The%20Effect%20Of%20Lersivirine%20On%20The%20Pharmacokinetics%20Of%20S-%20And%20R-Methadone